CLINICAL TRIAL: NCT01682889
Title: The Effect of High Dose Arginine Infusion on Hemodynamic and Peripheral Microcirculation: a Randomized, Controlled Clinical Trial in Patients Receiving Peripheral Vascular Surgery
Brief Title: The Effect of High Dose Arginine Infusion on Hemodynamic and Peripheral Microcirculation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical Scientific Fund of the Mayor of Vienna (Other)
Responsible Party: Principal Investigator, Ass.-Prof. DI Dr. Barbara Wessner, Ass.-Prof. DI Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MUW_Arginin
Record Dates: First submitted 2012-09-03; First posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): NaCl 0.9% intravenously for 24 hours after induction of anaesthesia
  Interventions: Dietary Supplement: Placebo
- Arginine (Active Comparator): L-arginine-hydrochlorid (0.35 g/kg body weight) intravenously for 24 hours after induction of anaesthesia
  Interventions: Dietary Supplement: Arginine

INTERVENTIONS:
Dietary Supplement: Arginine — L-arginine-hydrochlorid (0.35 g/kg body weight) intravenously for 24 hours
  Arms: Arginine
Dietary Supplement: Placebo — NaCl 0.9% intravenously for 24h
  Arms: Placebo

SUMMARY:
The aim of this study was to investigate the effect of a 24- hrs L-arginine infusion on hemodynamic and on parameters of microcirculation in patients with peripheral arterial occlusive disease (PAOD).

ELIGIBILITY:
Inclusion Criteria:

* female or male patients receiving peripheral bypass surgery
* age between 55 and 75 years

Exclusion Criteria:

* metabolic acidosis

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in temperature gradient at 3h post-surgery | baseline and 3h post-surgery
  One temperature probe is attached to the index finger of the lying patients, a second probe at the radial side of the forearm, midway between elbow and the wrist. Temperature gradient is calculated by subtracting the value obtained at the fingertip from the forearm value and expressed in °C.

SECONDARY OUTCOMES:
Change from baseline in Laser Doppler blood perfusion imaging at 1h | baseline & 1h post-surgery
  Perfusion values are expressed as arbitrary perfusion units.
Change from baseline in Laser Doppler blood perfusion imaging at 2h | baseline & 2h post-surgery
  Perfusion values are expressed as arbitrary perfusion units.
Change from baseline in Laser Doppler blood perfusion imaging at 3h | baseline & 3h post-surgery
  Perfusion values are expressed as arbitrary perfusion units.
Change from baseline in Laser Doppler blood perfusion imaging at 24h | baseline & 24h post-surgery
  Perfusion values are expressed as arbitrary perfusion units.
Change from baseline in Laser Doppler blood perfusion imaging at 48h | baseline & 48h post-surgery
  Perfusion values are expressed as arbitrary perfusion units.
Change from baseline in asymmetric dimethylarginine (ADMA) at 3h | baseline & 3h post-surgery
  Asymmetric dimethylarginine is measured by ELISA and expressed in µmol/l.
Change from baseline in asymmetric dimethylarginine (ADMA) at 24h | baseline & 24h post-surgery
  Asymmetric dimethylarginine is measured by ELISA and expressed in µmol/l.
Change from baseline in asymmetric dimethylarginine (ADMA) at 48h | baseline & 48h post-surgery
  Asymmetric dimethylarginine is measured by ELISA and expressed in µmol/l.
Change from baseline in plasma arginine concentration at 3h | baseline & 3h post-surgery
  L-arginine concentration is measured by HPLC and expressed in µmol/l.
Change from baseline in plasma arginine concentration at 24h | baseline & 24h post-surgery
  L-arginine concentration is measured by HPLC and expressed in µmol/l.
Change from baseline in plasma arginine concentration at 48h | baseline & 48h post-surgery
  L-arginine concentration is measured by HPLC and expressed in µmol/l.
Change from baseline in temperature gradient at 1h | baseline & 1h post-surgery
  One temperature probe is attached to the index finger of the lying patients, a second probe at the radial side of the forearm, midway between elbow and the wrist. Temperature gradient is calculated by subtracting the value obtained at the fingertip from the forearm value and expressed in °C.
Change from baseline in temperature gradient at 2h | baseline & 2h post-surgery
  One temperature probe is attached to the index finger of the lying patients, a second probe at the radial side of the forearm, midway between elbow and the wrist. Temperature gradient is calculated by subtracting the value obtained at the fingertip from the forearm value and expressed in °C.
Change from baseline in temperature gradient at 24h | baseline & 24h post-surgery
  One temperature probe is attached to the index finger of the lying patients, a second probe at the radial side of the forearm, midway between elbow and the wrist. Temperature gradient is calculated by subtracting the value obtained at the fingertip from the forearm value and expressed in °C.
Change from baseline in temperature gradient at 48h | baseline & 48h post-surgery
  One temperature probe is attached to the index finger of the lying patients, a second probe at the radial side of the forearm, midway between elbow and the wrist. Temperature gradient is calculated by subtracting the value obtained at the fingertip from the forearm value and expressed in °C.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Michael Hiesmayr, Prof. Dr., Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria